CLINICAL TRIAL: NCT04227340
Title: Prevention of Oral Mucositis in Children and Adolescents Undergoing Hematopoietic Stem Cell Transplant Using Photobiomodulation Therapy
Brief Title: Prevention of Oral Mucositis Using Photobiomodulation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Association of Pediatric Hematology Oncology Nurses (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PrOM; NCI-2020-00101 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Results first posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Oral Mucositis
Keywords: Adolescents; Autologous Transplant; Chemotherapy; Children; Extra-oral Photobiomodulation Therapy; HCT; Hematopoietic Stem Cell Transplant; Low Level Light therapy; Oral Mucositis; PBM; Photobiomodulation Therapy
MeSH Terms: conditions — Stomatitis | interventions — Low-Level Light Therapy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Photobiomodulation Therapy (PBM) (Experimental): The PBM will be administered extra-oral and intra-oral.
  Interventions: Device: Photobiomodulation Therapy (PBM); Other: Pain and Oral Function Assessment; Other: Parent-Reported Satisfaction Survey

INTERVENTIONS:
Device: Photobiomodulation Therapy (PBM) — The PBM will be delivered through application of the LED Cluster Probe externally to the right external buccal, left external buccal, mid face with mouth open and submandibular and left/right cervical. Patients who develop an oral lesion, intra-oral directed therapy will be administered with the dental light probe. For patients that can tolerate, an intraoral probe will deliver light directly onto the oral mucosa, this will then replace the mid face application with mouth open. Each laser application will be timed at 60 seconds.
  Other Names: THOR 69 diode LED cluster probe (1390mW); PBM therapy
Other: Pain and Oral Function Assessment — After the 6-minute laser/ treatment session the child and parent will complete the mucositis evaluation scale on paper or ipad which includes self-report oral function specific to ability to swallow, eat and drink, as well as the patient's self-reported need for medication specific to mouth pain.
  Other Names: Mucositis Evaluation Scale
Other: Parent-Reported Satisfaction Survey — A parent-reported satisfaction survey will be administered via paper questionnaire after the initial LLLT treatment. Parent satisfaction will be reported by parents on a 5-point Likert scale to questions adapted from a parent satisfaction survey used in a study regarding child life services in pediatric imaging.
  Other Names: Survey

SUMMARY:
Oral mucositis is a significant and common toxicity experienced by patients who receive high-dose chemotherapy as a preparatory regimen for a hematopoietic cell transplant (HCT). Furthermore, oral mucositis has been reported as the single most debilitating side effect reported by patients undergoing HCT. The incidence of HCT mucositis among adults is estimated to range between 76% and 89%; however, comparisons are difficult due to variability in patient ages, treatments and criteria for scoring oral mucositis.

The use of intra-oral photobiomodulation (PBM) therapy in adult patients after the development of oral mucositis is well documented and now included in the international mucositis guidelines, with limited evidence in pediatrics. This study will build evidence for the incorporation of extra-oral PBM therapy into daily nursing care of children and adolescents undergoing HCT. This intervention has potential in providing evidence for efficacy in the prevention and treatment of oral mucositis, the single most debilitating side effect reported by patients undergoing HCT.

Primary Objective:

* To evaluate feasibility and efficacy of photobiomodulation therapy (PBM) in reducing oral mucositis in children and adolescents at risk for grade 3 oral mucositis undergoing an allogeneic hematopoietic cell transplant (HCT).

Secondary Objective:

* To compare clinical manifestations associated with the development of oral mucositis between those treated with daily PBM and a matched control. Clinical factors to include: grade and duration or oral mucositis.

Exploratory Objective:

* To evaluate efficacy of photobiomodulation therapy in autologous patients at risk for grade 3 oral mucositis compared to matched control.
* To evaluate utilization of play-based procedural preparation and treatment feasibility and parental satisfaction.

DETAILED DESCRIPTION:
Children, adolescents and young adults admitted for an allogeneic HCT and those determined by the transplant team to be at risk for grade 3 oral mucositis will be eligible to receive PBM (34 x 660nm 10mW, 35 x 850nm 30mW: 1390 mW total power output) at an irradiance of 50mW/cm2. The PBM treatment will be administered via the THOR Model LX2M unit.

After low light therapy consent, participants will be offered the opportunity to receive a play-based preparation. Those who elect to receive this child life preparation will be scheduled to meet with a trained certified child life specialist (CCL) prior to admission. The play-based preparation will incorporate age and developmentally appropriate explanations of the non-invasive procedure and will be adapted to each patient's psychosocial and cognitive developmental needs.

Observation and treatment will begin the first day of conditioning (plus/minus 2 days). Those undergoing an allogeneic HCT will have treatment daily until Day +20 or engraftment (ANC ≥ 500 for two consecutive days). For those undergoing an autologous transplant, treatment will continue until engraftment (ANC ≥ 500 for two consecutive days) or until the patient is without mucositis for two consecutive days.

The PBM will be administered extra-oral and intra-oral by trained research staff. Direct aim of the laser into the eye will be avoided and safety spectacles will be used with laser therapy. The safety spectacles will be prescribed according to age, with the adjustable Ibis Infant eye protection for patients less than 1 year of age and the adjustable kids laser safety googles for the young child. Patients, staff, and observers will wear laser safety glasses while PBM is in use.

The parent may hold the device in place with assistance from the trained persons. After the initial LLLT treatment, a parent-reported satisfaction survey will be administered via paper questionnaire.

The observation of oral mucositis will be conducted by non-study staff and conducted as clinical care by the nurse, advanced practice provider and/or physician. Each patient will have a daily oral assessment, with documentation of mucositis, grade, duration, pain assessment, days of nutrition support, use of narcotics, positive oral and blood cultures. All patients will receive the standard mouth care regimen prescribed for transplant patients.

Each patient will be matched and compared to a previously treated patient. The comparison will be matched on primary disease, conditioning regimen, age and sex, with comparison of treatment variables of mucositis grade, duration, pain medications, days of nutritional support, blood and oral cultures, to day +20 or engraftment (depending upon which occurs first).

ELIGIBILITY:
Inclusion Criteria:

* No age limitation
* To be admitted for an allogeneic hematopoietic cell transplant
* All eligible autologous hematopoietic cell transplant, at risk for grade 3 mucositis per transplant service secondary to conditioning regimen or previous history of grade 3 mucositis
* Dental exam prior to admission, as per preadmission criteria
* Willingness of research participant to provide assent/consent and parent/ legal guardian/representative to give written informed consent.

Exclusion Criteria:

* Deemed by transplant team as unable to participate
* Known sensitivity to light therapy
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* CAR-Tcell Protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Mandrell, PhD, RN, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 patients were enrolled between February 2020 and May 2021
  Historical Matched Controls were not enrolled on this study, therefore; they are not included in the protocol enrollment number.
Pre-assignment Details: Forty-three (43) participants were enrolled with 3 participants withdrawing consent prior to the start of treatment.
  Historical Matched Controls: Information obtained through chart reviews; matched on age, sex, primary diagnosis, and conditioning regimens; mucositis grade collected; previously treated on Bone Marrow transplant studies and non-protocol treatment plans (NPTP): 12 on NPTP; 2 on NCT01807611; 9 on NCT03849651; 17 on NCT02790515; not treated with Photobiomodulation.
Groups:
- Photobiomodulation Therapy (PBM): Acute Lymphoblastic Leukemia (ALL) and Acute Myeloid Leukemia (AML) patients undergoing Allogeneic transplant treated with Photobiomodulation
Period: Overall Study
Arm/Group | Photobiomodulation Therapy (PBM)
Started | 43
Completed | 40
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: The Historical Matched Controls were not enrolled on this study, therefore; they are not included in the protocol enrollment number.
Groups:
- Historical Matched Controls: Historical control matched: Patients matched on age, sex, primary diagnosis, conditioning regimen who were previously treated on Bone Marrow transplant studies and non-protocol treatment plans. Information was obtained through chart reviews.
- Total: Total of all reporting groups
Arm/Group | Photobiomodulation Therapy (PBM) | Historical Matched Controls | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (5.8) | 9.9 (5.3) | 10.4 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 21 | 22 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30 | 26 | 56
  Black | 6 | 8 | 14
  Asian | 1 | 1 | 2
  American Indian/Alaskan/White | 1 | 3 | 4
  Not Otherwise Specified | 2 | 2 | 4
Conditioning Regimen (choice=Chemotherapy) [Count of Participants; unit: Participants]
  Yes | 40 | 40 | 80
  No | 0 | 0 | 0
Conditioning Regimen (choice=Radiation) [Count of Participants; unit: Participants]
  No | 36 | 36 | 72
  Yes | 4 | 4 | 8
Primary Disease [Count of Participants; unit: Participants]
  Acute Lymphoblastic Leukemia (ALL) | 12 | 17 | 29
  Acute Myeloid Leukemia (AML) | 27 | 23 | 50
  Chronic Myeloid Leukemia (CML) | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Photo Biomodulation Therapy (PBM) in Reducing Oral Mucositis (OM) in Children and Adolescents at Risk for Grade 3 OM Undergoing an Allogeneic Hematopoietic Cell Transplant (HCT).
Description: Feasibility was assessed through the number of successful treatments (957) administered by the total number of attempted treatments (1023), providing the percentage of successful treatment administered. Daily treatment included 6 sites of PBM application, with application documented as receiving all 6 applications, in part treatment (at least one to five sites) or no treatment. A successful treatment was defined as successfully administered to 4 or more sites. Reasons for partial or no treatment was documented. Criteria for feasibility was 75%.
Time Frame: Daily assessment from day 1 of conditioning to 20 days after transplant or engraftment (2 consecutive days of an Absolute Neutrophil Count (ANC)>500)
Population: All PrOM study patients who received allogeneic transplant. Forty participants were treated daily for a total of 1023 patient encounters, during 66 patient encounters we were unable to treat 4 or more sites
Measure: Number (95% Confidence Interval); unit: percentage of successful treatments
Units Other Than Participants: Treatment Encounters
Arm/Group | Photobiomodulation Therapy (PBM)
Number analyzed (Participants) | 40
Number analyzed (Treatment Encounters) | 1023
percentage of successful treatments | 93 [93 to 94]

2. Primary Outcome: Efficacy of Photo Biomodulation Therapy (PBM) in Reducing Oral Mucositis (OM) in Children and Adolescents at Risk for Grade 3 OM Undergoing an Allogeneic Hematopoietic Cell Transplant (HCT).
Description: It was estimated from a retrospective review of HCT patients that 71% of participants undergoing a HCT developed grade 3 mucositis. With an estimated clinically meaningful effect size of 20% for PBM, the estimated percentage of PBM participant to develop grade 3 mucositis was set at 51%. An interim analysis was conducted after the enrollment of 40 participants.
Time Frame: as for outcome 1
Population: All patients who received at least 75% of the attempted PMB(n=40).
Measure: Count of Participants; unit: Participants
Groups:
- Photobiomodulation Treated: Acute Lymphoblastic Leukemia (ALL) and Acute Myeloid Leukemia (AML) patients undergoing Allogeneic transplant treated with Photobiomodulation
Arm/Group | Photobiomodulation Treated
Number analyzed (Participants) | 40
Participants | 8
Statistical Analysis 1: Comparison: Photobiomodulation Treated; The count, percentage and confidence interval were calculated for allogeneic HCT participants who receive PBM and developed Grade 3 mucositis. Whether the percentage of the prospective sample is significantly different from the estimated rate of 71% was accessed; Test type: Other — The count, percentage and confidence interval will be calculated for allogeneic HCT patients who receive PBM and develop Grade 3 mucositis; Odds Ratio (OR) = 0.2, 95% CI 2-sided [0.091 to 0.356] — Odds of grade 3 in Allogeneic group compared to historical rates. The study efficacy of mucositis reduction by 20% with an estimation of 51% developing grade 3 mucositis

3. Secondary Outcome: Assess the Severity of Mucositis Grade 1-3 and Duration for Each Patient Treated With PBM Compared to Matched Controls
Description: Patients were ranked according to the severity of their mucositis (a weighted average of mucositis intensity (grade 1-3) by number of days duration)
Time Frame: as for outcome 1
Population: Within each grade of mucositis (1-3) participants and controls were ranked against each other by days of mucositis duration. Each participant and control had 3 rankings for the 3 mucositis grades. The weighted average for each participant and control was calculated. Within each group (participant vs. control) there was a ranking (1-35 with the lower score being more severe mucositis). Statistical analysis then compared the weighted average between the two groups.
Measure: Number; unit: Days of mucositis within each grade
Arm/Group | Photobiomodulation Treated | Historical Matched Controls
Number analyzed (Participants) | 40 | 40
Days of mucositis within each grade
  Grade 1 | 143 | 177
  Grade 2 | 80 | 178
  Grade 3 | 19 | 46
Statistical Analysis 1: Comparison: Photobiomodulation Treated vs Historical Matched Controls; Test type: Superiority; p = 0.03, Wilcox Rank Sum

4. Secondary Outcome: Compare the Mucositis Grade and Duration Between Those Who Received PBM and Match Control.
Description: Participants treated with PBM therapy were matched to a transplant control who was not treated with PBM. Patients were matched by age, sex, primary disease and transplant conditioning regimen. Total days of grade 1 OM were calculated between PBM treated and untreated
Time Frame: as for outcome 1
Population: All patients in treatment and control group who developed grade 1 at various days, their duration of grade 1 data was used.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Overall: Photobiomodulation Treated:
  Acute Lymphoblastic Leukemia (ALL) and Acute Myeloid Leukemia (AML) patients undergoing Allogeneic transplant treated with Photobiomodulation
  Historical control matched: Patients matched on age, sex, primary diagnosis, conditioning regimen who were previously treated on Bone Marrow transplant studies and non-protocol treatment plans. Information was obtained through chart reviews.
Arm/Group | Photobiomodulation Treated | Historical Matched Controls | Overall
Number analyzed (Participants) | 40 | 40 | 80
Days | 3.58 (2.91) | 4.43 (3.85) | 4 (3.42)

5. Secondary Outcome: Compare the Mucositis Grade and Duration Between Those Who Received PBM and Match Control
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (Full Range); unit: Days
Arm/Group | Photobiomodulation Treated | Historical Matched Controls | Overall
Number analyzed (Participants) | 40 | 40 | 80
Days | 3 [0 to 10] | 4 [0 to 19] | 4 [0 to 19]
Statistical Analysis 1: Comparison: Photobiomodulation Treated vs Historical Matched Controls; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Compare the Mucositis Grade and Duration Between Those Who Received PBM and Match Control
Description: Participants treated with PBM therapy were matched to a transplant control who was not treated with PBM. Patients were matched by age, sex, primary disease and transplant conditioning regimen. Total days of grade 2 OM were calculated between PBM treated and untreated.
Time Frame: as for outcome 1
Population: All patients in treatment and control group who developed grade 2 at various days, their duration of grade 2 data was used.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Photobiomodulation Treated | Historical Matched Controls | Overall
Number analyzed (Participants) | 40 | 40 | 80
Days | 2 (2.10) | 4.45 (4.99) | 3.23 (4)

7. Secondary Outcome: Compare the Mucositis Grade and Duration Between Those Who Received PBM and Match Control
Description: as for outcome 6
Time Frame: as for outcome 1
Description (as registered): Participants treated with PBM therapy were matched to a transplant control who was not treated with PBM. Patients were matched by age, sex, primary disease and transplant conditioning regimen. Total days of grade 3 OM were calculated between PBM treated and untreated.
Population: as for outcome 6
Measure: Median (Full Range); unit: Days
Arm/Group | Photobiomodulation Treated | Historical Matched Controls | Overall
Number analyzed (Participants) | 40 | 40 | 80
Days | 1.5 [0 to 6] | 2.5 [0 to 16] | 2 [0 to 16]
Statistical Analysis 1: Comparison: Photobiomodulation Treated vs Historical Matched Controls; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Compare the Mucositis Grade and Duration Between Those Who Received PBM and Match Control.
Description: Participants treated with PBM therapy were matched to a transplant control who was not treated with PBM. Patients were matched by age, sex, primary disease and transplant conditioning regimen. Total days of grade 3 OM were calculated between PBM treated and untreated.
Time Frame: as for outcome 1
Population: All patients in treatment and control group who developed grade 3 at various days, their duration of grade 3 data was used.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Photobiomodulation Treated | Historical Matched Controls | Overall
Number analyzed (Participants) | 40 | 40 | 80
Days | 0.47 (1.15) | 1.15 (2.18) | 0.81 (1.77)

9. Secondary Outcome: Compare the Mucositis Grade and Duration Between Those Who Received PBM and Match Control
Description: as for outcome 8
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Median (Full Range); unit: Days
Arm/Group | Photobiomodulation Treated | Historical Matched Controls | Overall
Number analyzed (Participants) | 40 | 40 | 80
Days | 0 [0 to 5] | 0 [0 to 8] | 0 [0 to 8]
Statistical Analysis 1: Comparison: Photobiomodulation Treated vs Historical Matched Controls; Test type: Superiority; p = 0.1, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Days of Hospitalization Between Groups
Description: Total days of hospitalization between the treated and control group
Time Frame: From the time of admission to discharge
Population: All patients in treatment and control group during their hospitalization for Bone Marrow Transplant (BMT).
Measure: Mean (Standard Deviation); unit: Days of hospitalization
Arm/Group | Photobiomodulation Treated | Historical Matched Controls
Number analyzed (Participants) | 40 | 40
Days of hospitalization | 32.4 (6.40) | 40.2 (15.7)

11. Secondary Outcome: Days of Hospitalization Between Groups
Description: Total days of hospitalization between the treated and control group
Time Frame: From the time of admission to discharge
Population: All patients in treatment and control group during their hospitalization for BMT.
Measure: Median (Full Range); unit: Days of hospitalization
Arm/Group | Photobiomodulation Treated | Historical Matched Controls
Number analyzed (Participants) | 40 | 40
Days of hospitalization | 32 [23 to 49] | 35 [23 to 105]
Statistical Analysis 1: Comparison: Photobiomodulation Treated vs Historical Matched Controls; Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events associated with PBM will be monitored daily from day 1 of conditioning to 20 days after transplant, or engraftment which is defined as 2 consecutive days of an Absolute Neutrophil Count (ANC)>500. The control group was not enrolled on this study, therefore; adverse events were not monitored/assessed.
Arm/Group | Photobiomodulation Therapy (PBM)
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT04227340/Prot_SAP_001.pdf
  • Informed Consent Form (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT04227340/ICF_000.pdf